CLINICAL TRIAL: NCT05055453
Title: ESolutions Functions for Children and Young People With the myPhonak App
Brief Title: MyPhonak App Junior Pediatric Usability and Benefit Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-85, Sonova 2020_15
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental Study Group (Experimental): Participants age 8-17 with bilateral hearing loss will be fit with Phonak BTE hearing aids and given access to the Phonak hearing app. The participants will use the app to adjust the hearing aid microphone and noise reduction settings.
  Interventions: Device: MyPhonak Junior App; Device: Phonak Sky hearing aid

INTERVENTIONS:
Device: MyPhonak Junior App — The app is an accessory to the hearing aids which allows the user to make adjustments to their hearing aid in real-time. The hearing aid does not require the use of the app, but the objective of this study is to evaluate the effects of the user adjustments made via the app on the participant's speech intelligibility with the hearing aid.
Device: Phonak Sky hearing aid — A Behind-The-Ear hearing aid (BTE) fit to hearing impaired persons with mild to severe hearing loss.

SUMMARY:
Participants age 8-17 with bilateral hearing loss will be fit with Phonak BTE (Behind-The-Ear) hearing aids and given access to the myPhonak Junior hearing app. The participants will use the app to adjust the hearing aid microphone and noise reduction settings.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between the ages of 7 and 17 years old.
* bilateral mild to severe hearing loss
* experienced hearing aid users for 6+ months

Exclusion Criteria:

* any additional disabilities to the hearing impairment
* inability to complete the study procedures

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Läßig, M.D, M.D., Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Universitätsmedizin Mainz, HNO-Klinik, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Study Group
Started | 16
Completed | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Study Group
Number analyzed (Participants) | 16
Age, Customized [Median (Full Range); unit: years] | 12 [8 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 16

OUTCOME MEASURES:

1. Primary Outcome: dB SNR (Decibel Signal to Noise Ratio) Score Using the OLSA (Oldenburg Sentence Test) Speech in Noise Test
Description: Target speech is presented from a speaker in front of participant while background noise is presented from 4 surrounding speakers. The level of noise is presented at 65 dB SPL (Sound Pressure Level),with target speech presented at variable levels, both louder and softer than the noise. The dB SNR is the level at which the participant can correctly repeat 50% of the words. A lower/negative dB SNR is better, indicating that 50% of the speech is understood when noise is louder than or close to the level of speech. This test was given in three, randomized conditions for each participant at two visits: 1) hearing aids in Automatic, 2) hearing aids in Automatic but Directionality and Noise Reduction customized by participant using the app (i.e. "preferred" settings), and 3) hearing aids in Automatic but with the Directionality set to lowest level 0, (i.e. omnidirectional), and Noise Reduction set to the highest level 10,or all the way on (i.e., "extreme").Results of both visits was averaged
Time Frame: Day 1 of study, repeated on Day 14 of study
Population: All participants who completed the testing for at least one clinic visit.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Experimental Study Group
Number analyzed (Participants) | 16
dB
  dB SNR for Automatic program, both visits averaged | -1.33 (3.93)
  dB SNR for preferred settings of volume, NR, and Directionality, both visits averaged | -2.83 (3.37)
  dB SNR for extreme setting, both visits averaged | 0.08 (4.15)
Statistical Analysis 1: Comparison: Experimental Study Group; Test type: Other — A Shapiro Wilks test was used to test for normal distribution of the data; p < 0.001, Durbin-Conover Pairwise Comparison — Result for comparison between automatic only and "preferred" app settings
Statistical Analysis 2: Comparison: Experimental Study Group; A Shapiro Wilks test was used to test for normal distribution of the data; Test type: Other; p < 0.001, Durbin-Conover Pairwise Comparison — Result of comparison between "preferred" app setting and "extreme" app setting
Statistical Analysis 3: Comparison: Experimental Study Group; A Shapiro Wilks test was used to test for normal distribution of the data; Test type: Other — Result of comparison between automatic only and "extreme" app setting; p = 0.002, Durbin-Conover Pairwise Comparison

2. Secondary Outcome: Assessment of Hearing Situations in Children's Every Day Lives Questionnaire
Description: A German-language questionnaire which asks student to rate their listening quality in different environments. Participants compared their listening quality with hearing aids alone versus hearing aids plus the app. Rating scale is from 1 to 5 with 1 = mostly easy and 5 = mostly difficult, so a lower score is better, however a rating of 0 = no change. Participants were given one copy of questionnaire to fill out during week 1 of home trial, and a second copy to fill out during week 2 of home trial. Results are reported separately for week 1 and week 2.
Time Frame: Completion of first home trial at day 7, and completion of second home trial at day 14
Population: All participants who completed at least one home trial and one questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Study Group
Number analyzed (Participants) | 15
score on a scale
  Rating of listening quality Hearing Aid only first home trial | 2.61 (1.36)
  Average rating of listening quality Hearing Aid with app adjustments first home trial | 1.88 (1.16)
  Rating of listening quality Hearing Aid only second home trial | 2.42 (1.54)
  Rating of listening quality Hearing Aid with app adjustments second home trial | 1.55 (1.05)
Statistical Analysis 1: Comparison: Experimental Study Group; Test type: Other — Analysis of first home trial; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Experimental Study Group; Analysis of second home trial; Test type: Other; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Experimental Study Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05055453/Prot_SAP_000.pdf